CLINICAL TRIAL: NCT04259541
Title: Selected Aspects of Mental Health of Athletes
Status: Completed | Type: Observational
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Masa Cernelic Bizjak, Principal investigator, University of Primorska
Other Study IDs: UPrimorska
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Mental Health Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Psychodiagnostic — Intensity and frequency of specific symptoms, signs of problems in mental health

SUMMARY:
The study will assess the prevalence of mental health problems among different athletes. The study is based on the application of the battery of psychodiagnostic questionnaires, which were chosen aiming at investigating the prevalence of different symptoms related to problems in mental health or disorders.

This descriptive cross-sectional study will undertake sample with athletes categorized by the quality of their achievement.

DETAILED DESCRIPTION:
In the field of sports, there is a lot of knowledge about sports injuries, nutrition and regeneration. Much less is known about mental health among athletes. The investigators often think that the incidence of mental problems is low among top athletes. As the main cause of this misconception, the authors attribute the idealization of sports and athletes. Both the professional and the lay public are often of the opinion that only mentally strong individuals can be successful, which of course means that there is no place in the highest level for individuals with mental problems and disorders.

The clinical study will be performed with 400-500 athletes of both genders aged 18 to 40, from Slovenia. The investigators will invite all athletes who have been categorized in the current year and classified into the membership category, i.e. national, international, world or Olympic class (there were 500 at the last categorization) and they compete in various sports disciplines. The study will be designed as a cross-sectional study. For the purpose of the research, the investigators will use a battery of psychodiagnostic questionnaires consisting of five parts: demographics and sport characteristic, depression symptomatic, anxiety symptomatic, eating problems, alcohol use and abuse and resilience characteristics of individual athlete.

ELIGIBILITY:
Inclusion Criteria:

* Included in competitive play
* Is a professional athlete or participates in organized professional sports activities

Exclusion Criteria:

* Present injuries
* Recreational athletes
* Any other significant diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Atletes at a competitive level, coming from different sports.
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Intensity and frequency of specific symptoms | Baseline
  Intensity and frequency of specific symptoms could be the signs of problems in mental health

SECONDARY OUTCOMES:
Depressive symptomatology | Baseline
  The degree of depressive symptomatology (physical, affective, cognitive and behavioral symptoms) will be measured with The Depression Scale Center
Pathological eating patterns | Baseline
  The degree of pathological eating patterns will be measured with Eating Attitude Test Questionnaire (EAT-26; Garner and Garfinkel, 1979) as high levels of preoccupation with diet, weight, and other pathological eating patterns.
Level of risky alcohol consumption | Baseline
  Alcohol Use Disorders Identification Test (AUDIT); World Health Organization 2001 The level of risky alcohol consumption will be assessed with a questionnaire (designed by the World Health Organization) that defines the type of consumption and the level of risk of drinking alcohol.
Resilience | Baseline
  The degree of personality resilience to fight the stress will be measured with Resilience Scale II -DRS II; Sinclair, Celina & Oliver, 2003).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of health care, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No
Group participant data will be available to other researchers.